CLINICAL TRIAL: NCT02484196
Title: Dyspareunia in Women With Endometriosis: Impact of Surgery on Sexual Health
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Other Study IDs: ENDODISP14
Record Dates: First submitted 2015-06-23; First posted 2015-06-29 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Dyspareunia; Endometriosis
MeSH Terms: conditions — Dyspareunia; Endometriosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Couples: Women, with their partners, referred to the Obstetrics and Gynecological Department of the University Hospital for surgical treatment of endometriosis.
  Interventions: Behavioral: Questionnaires
- Women: Women referred to the Obstetrics and Gynecological Department of the University Hospital for surgical treatment of endometriosis.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires

SUMMARY:
Endometriosis is a disease that affects different areas of individual functioning, including the area of sexual life. Women with endometriosis have an impairment of desire and sexual arousal, orgasmic capacity reducted because of the pain and deep dyspareunia. The aim of the study is to evaluate the effectiveness of surgery on dyspareunia in women with endometriosis, taking into account other variables involved in determining dyspareunia: the quality of the couple relationship, anxiety and depression, body image, coping strategies and resilience.

ELIGIBILITY:
Inclusion Criteria:

* Women affected by endometriosis with dyspareunia;
* Women in waiting list for surgery

Exclusion Criteria:

* Severe underlying comorbidities (gynecological, cardiovascular, respiratory, renal, hematological, endocrine, hepatic, gastrointestinal, neurological)
* Psychiatric diseases
* Refusal or inability to sign the informed consent
* Pregnancy
* Previous gynecological surgery
* End of couple relationship

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women, and their parteners, affected by endometriosis with dyspareunia, referred to the Obstetrics and Gynecological Department of the University Hospital for the treatment of endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Quality of sexual life | Cases were administered and fulfilled the questionnaires at the moment of diagnosis of endometriosis up to 4weeks; Change from baseline were evalueted 2 months after surgery